CLINICAL TRIAL: NCT07313501
Title: Evaluation of the PERC Score and the YEARS Algorithm in the Diagnosis of Pulmonary Embolism in the Emergency Department: a Retrospective Observational Study in the Emergency Department of the Strasbourg University Hospital
Brief Title: Evaluation of the PERC Score and the YEARS Algorithm in the Diagnosis of Pulmonary Embolism in the Emergency Department
Acronym: EP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9611
Record Dates: First submitted 2025-12-17; First posted 2026-01-02 (Actual); Last update posted 2026-01-02 (Actual); Status verified 2025-12

CONDITIONS: Pulmonary Embolism
Keywords: Pulmonary Embolism; PERC score; D-dimer testing; Chest CT angiography
MeSH Terms: conditions — Pulmonary Embolism

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The current diagnostic strategy for pulmonary embolism relies on clinical evaluation, followed by D-dimer testing and chest CT angiography. However, this approach leads to overuse of CT angiography. Diagnosis remains complex, with nonspecific clinical signs. Recent studies have explored new algorithms, such as the YEARS algorithm and the PERC score, which aim to support the diagnosis and reduce the need for imaging examinations. Their use could decrease waiting times in the emergency department and limit the need for additional investigations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patient (≥18 years)
* Patient admitted to the adult emergency department of the Strasbourg University Hospital over a 6-month period (January to June 2024), for whom a D-dimer test and chest imaging (thoracic CT angiography or ventilation/perfusion scintigraphy) were performed

Exclusion Criteria:

- No D-dimer test or test performed for another indication, no chest imaging (CT angiography or scintigraphy), long-term anticoagulant treatment.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: - Adult patient (≥18 years) admitted to the adult emergency department of the Strasbourg University Hospital over a 6-month period (January to June 2024), for whom a D-dimer test and chest imaging (thoracic CT angiography or ventilation/perfusion scintigraphy) were performed
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2025-02-26 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Number of patients who would not have required imaging if the PERC score and YEARS algorithm criteria had been applied | Up to 12 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service d'Urgences Médico-Chirurgicales Adules - CHU de Strasbourg - France, Strasbourg, France